CLINICAL TRIAL: NCT05389683
Title: Assessment of Improvement in Food Sensitivity Related Symptoms on Employment of Personalized Elimination Diet
Brief Title: Effect of Personalized Elimination Diet on Food Sensitivity Related Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vibrant America Clinical Lab (Industry)
Responsible Party: Principal Investigator, Hari Krishnamurthy, Director - Biomedical Engineering, Vibrant America Clinical Lab
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB # 1-1586736-1
Record Dates: First submitted 2022-05-19; First posted 2022-05-25 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Food Sensitivity
Keywords: Food Sensitivity; Elimination diet
MeSH Terms: conditions — Food Intolerance | interventions — Elimination Diets

STUDY DESIGN:
Intervention Model Description: It is a single group study in which a single group of subjects will receive a single intervention and the outcomes will be assessed over time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Elimination Diet (Experimental): Participants will be suggested an 'Elimination diet' that will be devoid of the reaction-inducing foods and it shall be followed for 4 weeks.
  Interventions: Behavioral: Elimination Diet

INTERVENTIONS:
Behavioral: Elimination Diet — An 'elimination diet' devoid of the reaction-inducing foods will be suggested for 4 weeks.

SUMMARY:
The goal is to identify food sensitivity in patients and assess whether the avoidance of the reaction-inducing foods via an 'elimination diet' leads to improvement in patient symptoms and overall well-being.

DETAILED DESCRIPTION:
After seeking appropriate consent, patients' blood samples will be tested for the reactivity toward 262 foods using peptide and protein microarrays. Food protein extraction will be carried out in different solvents such as water and alcohol. The peptide microarrays will synthesize the entire food proteins as peptides in situ while the protein microarrays will test for water-soluble and alcohol-soluble fractions. Thus, food sensitivity testing will be carried out at 3 different levels including water-soluble proteins, alcohol-soluble proteins, and peptides. Patients' blood samples can be tested at all 3 levels or a combination of these. This decision lies at the discretion of the physician.

Based on the test results and as per the physician's recommendations, a suitable elimination diet will be suggested to the patient. Personalized diet suggestions for each patient will be made by the physician. The patient will follow the diet for 4 weeks and blood samples will be tested again on completion of the diet, using peptides and protein microarrays. Additionally, based on the physician's recommendations, the time duration for which a patient follows the personalized elimination diet can be modified.

The patients will periodically have to fill out diagnostic questionnaires which will help assess the changes in their food sensitivity-related symptoms. Changes in the blood biomarkers and improvement in symptoms will be monitored during the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 to 65 years.
* Patients suffering from food sensitivity symptoms
* Patients having Immunoglobulin G (IgG) and Immunoglobulin A (IgA)-mediated food reactions leading to food sensitivity
* Patients agreeing to follow the diet per testing
* Patients willing to provide an informed consent

Exclusion Criteria:

* Patients suffering from chronic medical conditions like cancer
* Pregnant subjects
* Patients who have recently used antibiotics
* Patients who have previously undergone treatments for food allergies/sensitivities
* Patients who have been assigned an elimination diet before
* Patients who are already following a restricted diet of any kind
* Patients unwilling/unable to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2024-02-24 (Actual); Study Completion 2024-02-24 (Actual)

PRIMARY OUTCOMES:
Improvement in blood biomarker profile | Baseline - 4 weeks
  The peptide and protein microarrays will be used to test patients' blood samples prior to and post-employment of the elimination diet, and changes in the blood biomarker profile will be monitored. Testing will be carried out at baseline and then after 4 weeks, on completion of the diet.
Improvement in severity of food sensitivity symptoms | Baseline; Week 1; Week 2; Week 3; Week 4
  Food Sensitivity - Symptom Severity Scale (FS - SSS) is a 16-item questionnaire that will assess the severity of the patient's food sensitivity-related symptoms. The scores range from 0 (none) to 5 (severe).

SECONDARY OUTCOMES:
Food Sensitivity - Quality of Life Questionnaire (FS-QoL) | Baseline; Week 4
  The FS-QoL is a 21-item measure assessing the degree to which Food Sensitivity-related symptoms interfere with a patient's quality of life. Each item is rated on a 5-point Likert scale.
Food sensitivity - Global Improvement Scale (FS-GIS) | Week 4
  The FS-GIS is a single-item assessment of overall Food Sensitivity symptoms and improvement. This questionnaire will be filled out by the physician to report the patient's response to the given intervention. It poses the question to the physician "Compared to the patient's condition during admission to the project [prior to intervention initiation], has the patient's food sensitivity-related symptoms been:" The physician can select: 1 = Substantially Improved, 2 = Moderately Improved, 3 = Slightly Improved, 4 = No change, 5 = Slightly Worse, 6 = Moderately Worse, 7 = Substantially Worse.

CONTACTS AND LOCATIONS:
Overall Officials: Hari K Krishnamurthy, M.S., Principal Investigator — PI
Locations (9):
- United States (9):
  - Hope Natural Health, Gilbert, Arizona
  - Inside Out Aesthetics, Scottsdale, Arizona
  - Vitality MD's, Scottsdale, Arizona
  - Mr. Hari Krishnamurthy, San Carlos, California
  - Vitality Health and Wellness, Miami Beach, Florida
  - Institute for Hormonal Balance, Orlando, Florida
  - One Agora Integrative Health, Bloomington, Minnesota
  - Turnpaugh Health and Wellness Center - Manheim, Manheim, Pennsylvania
  - Turnpaugh Health and Wellness Center - Mechanicsburg, Mechanicsburg, Pennsylvania

IPD SHARING:
Plan to Share IPD: No